CLINICAL TRIAL: NCT02178553
Title: Randomized Non-inferiority Trial of Continuous Thoracic Epidural Analgesia Versus Single Intercostal Nerve Block After Thoracotomy
Brief Title: Study of Exparel Versus Epidural for Pain Control After Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James D. Hannon, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-002940
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-11

CONDITIONS: Pain Following Thoracotomy Surgery
Keywords: Thoracotomy; Pain
MeSH Terms: conditions — Pain | interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural (Active Comparator): In the epidural catheter (TEC) group, a thoracic epidural catheter will be placed at the level of T6-T8 and advanced 5 cm into the epidural space and a 3 ml test dose of lidocaine 1.5% will be administered before the induction of general anesthesia. Patients will be excluded from the study if the catheter cannot be placed. A bolus dose of 0.5 mg hydromorphone plus 4.5 ml 0.125% bupivacaine will be administered before surgical incision. An epidural infusion of 0.075% bupivacaine and 10 mcg/ml hydromorphone, prepared by the hospital pharmacy, will be started intraoperatively at a rate of 5 ml/hr.
  Interventions: Drug: Epidural
- Intercostal bupivicaine (Exparel) (Active Comparator): In the intercostal block (ICB) group, liposomal bupivacaine 1.3% (4 ml) will injected by the surgeon under direct vision into the proximal intercostal space at the level of the thoracotomy and one interspace above and below. In addition, liposomal bupivacaine 1.3 % (4 ml) will be injected at each of the chest tube exit sites. Thus, a total of 20 ml liposomal bupivacaine 1.3% (260 mg) will be administered.
  Interventions: Drug: Intercostal Bupivicaine (Exparel)

INTERVENTIONS:
Drug: Epidural
  Arms: Epidural
Drug: Intercostal Bupivicaine (Exparel)
  Arms: Intercostal bupivicaine (Exparel)

SUMMARY:
Unilateral intercostal nerve blocks provide pain control as effectively as a continuous thoracic epidural, and will a lower incidence of side effects.

DETAILED DESCRIPTION:
In this study we will study to see if a single set of unilateral intercostal nerve blocks provides pain control as effectively as a continuous thoracic epidural, and will a lower incidence of side effects. Although the anesthesiologists involved in providing care for patients having thoracotomy incisions at St. Mary's Hospital are experts at placing thoracic epidural catheters, this study will attempt to show that a less technically challenging procedure done by surgeons intra-operatively can provide comparable pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Undergoing thoracotomy (lobectomy, segmentectomy, wedge resection or pneumonectomy).

Exclusion Criteria:

* Planned chest wall resection or abdominal incision and/or gastroesophageal surgery;
* Current enrollment in another post-thoracotomy analgesic research protocol; pre-existing pain syndrome (such as fibromyalgia, complex regional pain syndrome or postherpetic neuralgia in a thoracic distribution);
* Daily opioid therapy;
* Current gabapentin or pregabalin therapy;
* Allergy to any study medication; coagulation or infectious issues that would preclude epidural catheter placement;
* Severe psychological disorders or inability to understand the study protocol; -Prisoners or other institutionalized individuals;
* Severe hepatic, renal or cardiovascular disorders.
* Women who are pregnant will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Hannon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epidural | Intercostal Bupivicaine (Exparel)
Started | 53 | 49
Completed | 45 | 39
Not Completed | 8 | 10
Not completed — Did not proceed to open thoracotomy | 7 | 3
Not completed — Physician Decision | 0 | 4
Not completed — Technical problem with injection | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural | Intercostal Bupivicaine (Exparel) | Total
Number analyzed (Participants) | 45 | 39 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (12.5) | 62.1 (10.8) | 61.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 19 | 21 | 40
  Sex: Male | 26 | 18 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 43 | 39 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.5 (6.1) | 28.8 (7.4) | 29.2 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores With Cough on First Postoperative Day
Description: Pain with cough documented using the numerical rating scale pain scores (0-10)
Time Frame: In the morning (8 am) on first postoperative day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epidural | Intercostal Bupivicaine (Exparel)
Number analyzed (Participants) | 45 | 39
units on a scale | 6.1 (2.7) | 6.9 (2.4)
Statistical Analysis 1: Comparison: Epidural vs Intercostal Bupivicaine (Exparel); Test type: Non-Inferiority — We determined that a difference of 1 unit between groups would be the bound for non-inferiorty; p = 0.142, t-test, 2 sided; Confidence Interval = 1, 90% CI 2-sided [-0.1 to 1.8]

2. Primary Outcome: Pain Scores With Cough on the Second Postoperative Day
Description: Pain with cough documented using the numerical rating scale pain scores (0-10). Zero indicates no pain, and 10 indicates the worst pain one could imagine.
Time Frame: In the morning (8 am) on the second postoperative day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epidural | Intercostal Bupivicaine (Exparel)
Number analyzed (Participants) | 45 | 39
score on a scale | 5.2 (2.1) | 6.0 (1.9)
Statistical Analysis 1: Comparison: Epidural vs Intercostal Bupivicaine (Exparel); Test type: Non-Inferiority — We determined that a difference of 1 unit between groups would be the bound for non-inferiorty; p = 0.101, t-test, 2 sided; Confidence Interval = 1, 90% CI 2-sided [0.4 to 1.9]

3. Secondary Outcome: Pain Scores at Rest in the Morning on the First Postoperative Day
Description: NRS pain scores on a 0-10 scale at rest at 8 am on the first postoperative day. Zero indicates no pain, and 10 indicates the worst pain one could imagine.
Time Frame: Each morning for two days postoperative
Measure: Mean (Standard Deviation); unit: NRS pain score on a scale from 0-10
Arm/Group | Epidural | Intercostal Bupivicaine (Exparel)
Number analyzed (Participants) | 45 | 39
NRS pain score on a scale from 0-10 | 2.9 (2.0) | 4.0 (2.2)
Statistical Analysis 1: Comparison: Epidural vs Intercostal Bupivicaine (Exparel); Test type: Non-Inferiority — We determined that a difference of 1 unit between groups would be the bound for non-inferiorty; p = 0.014, t-test, 2 sided; Confidence Interval = 1, 90% CI 2-sided [0.4 to 1.9]

4. Secondary Outcome: Pain Scores at Rest on the Second Postoperative Day
Description: NRS pain scores on a 0-10 scale at rest in the morning on the second postoperative day. Zero indicates no pain, and 10 indicates the worst pain one could imagine.
Time Frame: Each morning for two days postoperative
Measure: Mean (Standard Deviation); unit: NRS pain scores on a scale from 0-10
Arm/Group | Epidural | Intercostal Bupivicaine (Exparel)
Number analyzed (Participants) | 45 | 39
NRS pain scores on a scale from 0-10 | 2.8 (1.9) | 3.2 (1.6)
Statistical Analysis 1: Comparison: Epidural vs Intercostal Bupivicaine (Exparel); Test type: Non-Inferiority — We determined that a difference of 1 unit between groups would be the bound for non-inferiorty; p = 0.375, t-test, 2 sided; Confidence Interval = 1, 90% CI 2-sided [-0.3 to 1.0]

ADVERSE EVENTS:
Time Frame: 3 months from the date of surgery
Groups:
- Epidural: In the epidural catheter (TEC) group, a thoracic epidural catheter will be placed at the level of T6-T8 and advanced 5 cm into the epidural space and a 3 ml test dose of lidocaine 1.5% will be administered before the induction of general anesthesia. Patients will be excluded from the study if the catheter cannot be placed. A bolus dose of 0.5 mg hydromorphone plus 4.5 ml 0.125% bupivacaine will be administered before surgical incision. An epidural infusion of 0.075% bupivacaine and 10 mcg/ml hydromorphone, prepared by the hospital pharmacy, will be started intraoperatively at a rate of 5 ml/hr.
  Epidural
- Intercostal Bupivicaine (Exparel): In the intercostal block (ICB) group, liposomal bupivacaine 1.3% (4 ml) will injected by the surgeon under direct vision into the proximal intercostal space at the level of the thoracotomy and one interspace above and below. In addition, liposomal bupivacaine 1.3 % (4 ml) will be injected at each of the chest tube exit sites. Thus, a total of 20 ml liposomal bupivacaine 1.3% (260 mg) will be administered.
  Intercostal Bupivicaine (Exparel)
Arm/Group | Epidural | Intercostal Bupivicaine (Exparel)
All-Cause Mortality (participants affected / at risk) | 1/46 | 3/39
Serious Adverse Events (participants affected / at risk) | 5/46 | 5/39
Other Adverse Events (participants affected / at risk) | 3/46 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epidural (N=46) | Intercostal Bupivicaine (Exparel) (N=39)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1 — Re-intubation and mechanical ventilation after surgery
Prolonged hospital stay (Surgical and medical procedures) | 1 | 1 — Prolongation of existing hospitalization
Pulmonary complications (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Brochopleural fistula, empyema, or pneumonia
Myocardial infarction (Cardiac disorders) | 0 | 1 — Acute myocardial infarction diagnosis during the study period
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epidural (N=46) | Intercostal Bupivicaine (Exparel) (N=39)
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 0 — Pruritis during hospitalization

LIMITATIONS AND CAVEATS:
The study was stopped before the target number of participants was achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT02178553/Prot_SAP_000.pdf